CLINICAL TRIAL: NCT02990611
Title: A National, Prospective, Non-Interventional Study (NIS) of Nivolumab (BMS-936558) Monotherapy or in Combination With Ipilimumab in Patients With Advanced (Unresectable or Metastatic) Melanoma and in Patients With Adjuvant Nivolumab Therapy
Brief Title: Observational Study of Nivolumab Monotherapy or in Combination With Ipilimumab in Participants With Advanced Melanoma and in Participants With Adjuvant Nivolumab Therapy
Acronym: NICO
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-654
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Nivolumab/Ipilimumab combination therapy: Participants who start a new systemic therapy with nivolumab/ipilimumab combination therapy for the first time
- Cohort 2: Nivolumab monotherapy: Participants who start a new systemic therapy with nivolumab monotherapy for the first time
- Cohort 3: Nivolumab adjuvant therapy: Participants who start adjuvant treatment with nivolumab after complete surgical tumor resection and no evidence of disease

SUMMARY:
The purpose of this study is to describe the safety and effectiveness of nivolumab treatment, either in monotherapy or in combination with ipilimumab, overall and according to various subgroups of interest, in participants with advanced melanoma and in participants with adjuvant nivolumab therapy.

ELIGIBILITY:
Inclusion Criteria:

For Cohort 1 and 2: (Recruitment ended by 02/20/2020)

* Advanced melanoma (Stage III/Stage IV)
* Histologically confirmed diagnosis
* Treatment decision for nivolumab monotherapy or nivolumab/ipilimumab combination therapy has already been taken

For Cohort 3: (Recruitment ended by 08/31/2020)

* Primary diagnosis of advanced melanoma after complete surgical tumor resection and no evidence of disease
* Treatment decision for adjuvant nivolumab therapy has already been taken

Exclusion Criteria:

For Cohort 1 and 2: (Recruitment ended by 02/20/2020)

* Current primary diagnosis of a cancer other than advanced melanoma, that requires systemic or other treatment or has not been treated curatively (as per discretion of the investigator)
* Previous treatment with nivolumab, for nivolumab monotherapy cohort only
* Current active participation in an interventional clinical trial

For Cohort 3: (Recruitment ended by 08/31/2020)

* Current diagnosis of persisting advanced melanoma or a cancer other than advanced melanoma that requires systemic or other treatment or has not been treated curatively (as per discretion of the investigator)
* Current active participation in an interventional clinical trial

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who are at least 18 years of age of the time of treatment decision with a primary diagnosis of advanced melanoma (histologically confirmed Stage III [unresectable] or Stage IV skin, ocular, or mucosal melanoma) and whose physician has already decided to initiate a treatment with nivolumab or nivolumab/ipilimumab for the first time for the treatment of melanoma, according to the label approved in Germany. Participants with a current primary diagnosis of a cancer other than advanced melanoma, participants currently included in an interventional clinical trial, or participants who have already received nivolumab in a prior line of therapy (for monotherapy arm) will all be excluded from this study. Adult participants in the adjuvant nivolumab treatment cohort will be enrolled after complete surgical resection and no evidence of disease after the treating physician has decided to initiate an adjuvant therapy with nivolumab according to the label approved in Germany.
Sampling Method: Probability Sample
Enrollment: 1087 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) of nivolumab/ipilimumab combination therapy | 5 years
Relapse free survival (RFS) of adjuvant nivolumab therapy | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) of nivolumab monotherapy | 5 years
Overall survival (OS) of nivolumab monotherapy or nivolumab/ipilimumab combination therapy, according to other subgroups of interest | 5 years
Progression-free survival (PFS) of nivolumab monotherapy or nivolumab/ipilimumab combination therapy | 5 years
Overall response rate (ORR) of nivolumab monotherapy or nivolumab/ipilimumab combination therapy | 5 years
Best overall response (BOR) of nivolumab monotherapy and of nivolumab/ipilimumab combination therapy | 5 years
Best overall response rate (BORR) of nivolumab monotherapy or nivolumab/ipilimumab combination therapy | 5 years
Duration of response of monotherapy and combination therapy | Up to 5 years
Distribution of sociodemographic characteristics: Age | 5 years
Distribution of sociodemographic characteristics: Gender | 5 years
Distribution of sociodemographic characteristics: BMI | 5 years
Distribution of clinical characteristics: Initial diagnosis of melanoma | 5 years
Distribution of clinical characteristics: Diagnosis of advanced melanoma | 5 years
Distribution of clinical characteristics: Duration of disease from date of initial melanoma diagnosis to initial treatment in study, or date of study entry (if untreated) | 5 years
Distribution of clinical characteristics: Surgery of complete tumor resection and no evidence of disease | 5 years
Distribution of clinical characteristics: Clinical code and staging melanoma subtypes | 5 years
Distribution of clinical characteristics: Comorbidities | 5 years
Distribution of clinical characteristics: Diagnostic procedures | 5 years
Distribution of clinical characteristics: Mutation status | 5 years
Distribution of clinical characteristics: Performance status as measured by Eastern Cancer Oncology Group (ECOG) scale | 5 years
Distribution of clinical characteristics: Medical history | 5 years
Distribution of clinical characteristics: Concomitant medication | 5 years
Distribution of clinical characteristics: History of cancer | 5 years
Distribution of clinical characteristics: Previous enrollment in an interventional study randomized controlled trials (RCTS) | 5 years
Distribution of treatment patterns: Type of treatment previously received | 5 years
Distribution of treatment patterns: Stage of melanoma | 5 years
Distribution of treatment patterns: Current treatment details | 5 years
European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ C-30) | 5 years
Incidence of adverse events (AEs) | 5 years
Severity of adverse events (AEs) | 5 years
Distribution of management of adverse events (AEs) | 5 years
Overall survival (OS) of adjuvant therapy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Essen, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html